CLINICAL TRIAL: NCT01839877
Title: Intra-arterial Hepatic Beads Loaded With Irinotecan With Concomitant Chemotherapy With FOLFOX in Patients With Colorectal Cancer With Unresectable Liver Metastases: a Phase II Multicenter Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 1201 DEBIRI
Record Dates: First submitted 2013-04-12; First posted 2013-04-25 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer With Non Resectable Hepatic Metastasis
Keywords: Metastatic colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIA DEBIRI + systemic FOLFOX (Experimental): Intra-arterial hepatic beads loaded with irinotecan with systemic FOLFOX
  Interventions: Drug: HIA DEBIRI + systemic FOLFOX

INTERVENTIONS:
Drug: HIA DEBIRI + systemic FOLFOX

SUMMARY:
Treatment of patients with colorectal cancer having liver metastases is currently based on systemic chemotherapy.

Triple therapy with 5FU, oxaliplatin and irinotecan intravenously was effective in terms of response and secondary resectability, however it is particularly toxic.

Hepatic intra-arterial chemotherapy (HIA) has been the subject of several studies. It has shown good efficacy with oxaliplatin and FUDR. However, the procedure is difficult to set up and reserved for experienced centers.

The objective of this protocol is to use a triple therapy based on 5FU and oxaliplatin associated to irinotecan which is administered by hepatic intra-arterial route, loaded onto microbeads (DEBIRI). Furthermore, the procedure for chemo-embolization DEBIRI is limited to 2 sessions, and therefore could be more easily generalized.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal adenocarcinoma,
* Liver metastases radiologically or histologically proven
* At least one measurable liver lesions by RECIST v1.1
* Age ≥ 18 years
* WHO Index < or = 2
* Life expectancy ≥ 3 months
* No extrahepatic disease except lung nodules if number < or = 3 and size < 10 mm each
* Healthy liver <60%
* Primary tumor resected or still in place
* No prior chemotherapy for metastases treatment (except a perioperative chemotherapy, if the last cycle was administered at least 12 months ago)
* Adjuvant chemotherapy after resection of the primary authorized if the last cycle was administered at least 12 months ago
* Normal hepatic function: total bilirubin ≤ 1.5 N; AST ≤ 5N; ALT ≤ 5N and PAL ≤ 5N
* TP ≥ 60%
* Adequate hematologic function: ANC ≥ 1500/mm3, platelets ≥ 100 000/mm3, Hb ≥ 9g/dl
* Good renal function: creatinine clearance ≥ 60 mL / min
* No cardiac dysfunction: no cardiovascular events in the last 6 months or no NYHA ≥ 2

Exclusion Criteria:

* Patient eligible for curative treatment (resection and / or radiofrequency ablation) by a multidisciplinary decision (including the opinion of a liver surgeon)
* Pregnant or lactating woman or patients of both sexes and of childbearing age not using adequate contraception
* History of cancer, except skin cancer (other than melanoma), carcinoma in situ of the cervix uteri treated curative. Other cancers treated with curative intent are permitted provided they did not relapse over the last 5 years
* Peripheral neuropathy
* Inflammatory Bowel Diseases
* Intestinal obstruction
* Chronic liver disease (viral, alcoholic or metabolic)
* Immune Deficiency Syndromes (history of transplantation, infection with HIV)
* Known to have contraindications to 5FU, oxaliplatin, folinic acid, irinotecan or to contrast products
* Patients with known contraindications against hepatic embolization procedures:

Presence of biliary-digestive anastomosis or biliary stent Cruoric or tumor thrombosis of the portal vein

* Patient who for psychological, social, family or geographical reasons could not be followed up regularly
* Legal disability (persons deprived of liberty or under guardianship)
* Patient is not affiliated to a social security scheme
* Participation in another concurrent study investigating the effect of treatment and this until 4 weeks after the end of the concurrent study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julien TAIEB, Pr, Principal Investigator — Fédération Francophone de Cancérologie Digestive
Locations (9):
- France (9):
  - Hopital Saint André, Bordeaux
  - CHU - Hôpital François Mitterand, Dijon
  - Hôpital Prive Jean Mermoz, Lyon
  - Centre Léon Berard, Lyon
  - Institut Paoli Calmette, Marseille
  - CHU de la TIMONE, Marseille
  - Hôpital Europeen G Pompidou, Paris
  - CHU Charles Nicolle, Rouen
  - Hôpital Rangueil, Toulouse

REFERENCES:
- [Result] Pernot S, Pellerin O, Artru P, Monterymard C, Smith D, Raoul JL, De La Fouchardiere C, Dahan L, Guimbaud R, Sefrioui D, Jouve JL, Lepage C, Tougeron D, Taieb J; for FFCD1201-DEBIRI investigators/Collaborators. Intra-arterial hepatic beads loaded with irinotecan (DEBIRI) with mFOLFOX6 in unresectable liver metastases from colorectal cancer: a Phase 2 study. Br J Cancer. 2020 Aug;123(4):518-524. doi: 10.1038/s41416-020-0917-4. Epub 2020 Jun 8. PMID 32507854

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty eight patients were included in the study between May 2013 and December 2016.
Groups:
- HIA DEBIRI + Systemic FOLFOX: Patients received induction chemotherapy with FOLFOX: oxaliplatin 85 mg/m2 as a 2-h infusion at day 1, leucovorin 400 mg/m2 as a 120-min infusion at day 1 followed by 5FU 400 mg/m2 bolus at day 1 and 2400 mg/m2 46-h continuous 5FU infusion, 1 cycle every 2 weeks. Patients received treatment with DC Bead LUMI™ 100-300 loaded with irinotecan 50 mg/ml, 1 vial per lobe and per treatment (meaning 1 vial in case of unilobar administration, and 2 vials in case of bilobar administration). Each treatment session was performed 48-72 h after a chemotherapy cycle. Treatment administration was performed using a unilateral femoral approach.
Period: Overall Study
Arm/Group | HIA DEBIRI + Systemic FOLFOX
Started | 58
Completed | 57
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Baseline population is on ITT population meaning all patients included excepted the patient wrongly included (beacuase of pancreatic metastases and not colorectal metastases)
Groups:
- HIA DEBIRI + Systemic FOLFOX: Intra-arterial hepatic beads loaded with irinotecan with systemic FOLFOX
  HIA DEBIRI + systemic FOLFOX
Arm/Group | HIA DEBIRI + Systemic FOLFOX
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.14 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 57

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at 9 Months
Description: The primary endpoint was to evaluate the rate of patients alive without progression at 9 months after the start of treatment. Events to be considered for the endpoint were:
  * Progression : defined as radiological progression according to RECIST V1.1 criteria, as assessed by the investigator.
  * Death Patients who progressed or died (from any cause) within 9 months of starting treatment were considered as failure for the primary endpoint. The first event which occured will be taken into accoun
Time Frame: at 9 months after inclusion
Population: Primary endpoint was on mITT population meaning all the patients included in the study with at least one radiological assessments within the 9 months following the inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | HIA DEBIRI + Systemic FOLFOX
Number analyzed (Participants) | 56
Participants
  Patients alive without any progression | 30
  Patients with progression or death | 26

2. Secondary Outcome: Overall Survival
Description: It was defined as the time interval between the date of inclusion and the date of death (whatever the cause). Patients lost to follow-up or alive at the time of analysis were censored at the date of last news.
Time Frame: up to 4 years after patient's inclusion
Population: Endpoint was analyzed on the ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HIA DEBIRI + Systemic FOLFOX
Number analyzed (Participants) | 57
months | 37.4 [25.7 to 45.8]

ADVERSE EVENTS:
Time Frame: Up to the end of treatment for each patient, up to 3 years After the end of the treatment, patients were followed-up only for the overall survival up to 4 years.
Arm/Group | HIA DEBIRI + Systemic FOLFOX
All-Cause Mortality (participants affected / at risk) | 31/57
Serious Adverse Events (participants affected / at risk) | 27/57
Other Adverse Events (participants affected / at risk) | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIA DEBIRI + Systemic FOLFOX (N=57)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Enteritis (Gastrointestinal disorders) | 2
Gastrointestinal toxicity (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 3
Pancreatitis acute (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chest pain (General disorders) | 2
General physical health deterioration (General disorders) | 1
Injection site extravasation (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 4
Cholecystitis (Hepatobiliary disorders) | 2
Clostridium difficile colitis (Infections and infestations) | 3
Escherichia bacteraemia (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Superinfection bacterial (Infections and infestations) | 1
Superinfection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Deshydratation (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Tumor obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Confusional state (Psychiatric disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIA DEBIRI + Systemic FOLFOX (N=57)
Alopecia (Skin and subcutaneous tissue disorders) | 14
Urinary retention (Renal and urinary disorders) | 5
Allergic reaction (Immune system disorders) | 3
Cephalgia (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 5
Neuropathy (Nervous system disorders) | 49
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 31
Abdominal pain (Gastrointestinal disorders) | 15
Mucositis (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 32
Pancreatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 17
Anemia (Blood and lymphatic system disorders) | 56
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Cholecystitis (Hepatobiliary disorders) | 5
Hepatalgia (Hepatobiliary disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Thromboembolic event (Vascular disorders) | 3
Hypertension (Vascular disorders) | 8
Urinary tractus infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 49
Aspartate aminotransferase increased (Investigations) | 49
Total Bilirubin increased (Investigations) | 11
Creatinine increased (Investigations) | 10
Gammaglutamyltransferase increased (Investigations) | 28
White blood cell count decreased (Investigations) | 12
Lymphocytes decreased (Investigations) | 14
Phosphatases alcalines increased (Investigations) | 47
Weight loss (Investigations) | 4
Platelets decreased (Investigations) | 36
Neutropenia (Investigations) | 36
Anorexia (Metabolism and nutrition disorders) | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 9
Hyperkaliemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 15
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypokaliemia (Metabolism and nutrition disorders) | 14
Hyponatremia (Metabolism and nutrition disorders) | 19
Fatigue (General disorders) | 43
Fever (General disorders) | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT01839877/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT01839877/SAP_001.pdf